CLINICAL TRIAL: NCT04708197
Title: Role of rTMS in Recovery of Chronic Post Stroke Aphasia
Brief Title: Effect of High Frequency Transcranial Magnetic Stimulation on Recovery of Chronic Post-Stroke Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haidy Elshebawy, lecturer of Neurology ,MD ,faculty of medicine ,Cairo University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shebawy12345
Record Dates: First submitted 2021-01-09; First posted 2021-01-13 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Post Stroke Aphasia
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- aphasic patients (Other): post stroke aphasic patients will receive 10 sessions of high frequency rTMS 3 times per week over the damaged hemisphere without language therapy
  Interventions: Device: rTMS (repetitive transcranial magnetic stimulation )

INTERVENTIONS:
Device: rTMS (repetitive transcranial magnetic stimulation ) — applying high frequency TMS over the damaged hemisphere in chronic post stroke aphasic patients

SUMMARY:
high frequency excitatory rTMS applied over the dominant hemisphere in chronic post stroke aphasic patients to help the restoration of function by the left hemisphere

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) has been used in many studies as a novel intervention to treat disorders associated with stroke, including paralysis or dysphagia, hemispatial neglect, pain, and aphasia. Number of studies have demonstrated that low-frequency rTMS over the unaffected hemisphere can be useful for enhancing recovery in aphasic patients.. It is expected that application of high-frequency (facilitatory) rTMS over the dominant speech area would have a beneficial effect on improving speech performance.

The aim of this study is to evaluate the effect of excitatory high frequency rTMS on recovery of aphasia in chronic aphasic patients due to cerebrovascular stroke. Twenty patients with post-stroke aphasia were enrolled in this study. Patients were selected from those attending the stroke clinic of Neurology department, Cairo University during the period from June 2020 to November 2020. The protocol of the study was approved by the ethical committee of the Department of Neurology, Faculty of Medicine, Cairo University. The aim and procedures of the study were explained and written consent forms were taken from all patients prior to participation.

The eligibility criteria were: chronic post stroke nonfluent aphasia due to first-ever ischemic stroke in the distribution of middle cerebral artery diagnosed clinically and documented by computed tomography or magnetic resonance imaging on the brain, right handedness, both sexes, age ranged from 33 to 66 years old, duration at least 4 months from stroke onset, patients not receiving speech therapy and educated at least 10 years of education.

Exclusion criteria were: aphasia due to head injury or neurological disease other than stroke, other clinical forms of aphasia, unstable cardiac dysrhythmia or cardiac pacemaker, unstable or critically ill patients, current or history of epilepsy, skull wounds and pregnant females. Also patients with severe grade of weakness which interfere with writing ability.

The severity of aphasia was assessed for every patient using the Aphasia Severity Rating Scale (ASRS). According to this scale, language deficits were recognized ranging from 0 to 5 points.Every patient was then assessed for linguistic deficits using Kasr El-Eini Arabic Aphasia test (KAAT), which is a simple, rapid, standardized, valid, and reliable bedside test for Egyptian patients, literate and illiterate.

Neuroimaging studies (computerized tomography (CT) and/or magnetic resonance imaging (MRI) of the brain) were done for all participants.

Treatment procedures:

Real rTMS was applied three times per week for 10 sessions. Fifty trains of 10-Hz stimulation, each lasting for 5 seconds with an intertrain interval of 15 seconds were given through a figure-of-8 coil (9-cm diameter loop) positioned over the left Broca's area of the affected hemisphere (25 trains over pars triangularis followed by 25 trains over pars opercularis.The intensity of stimulation was set at 80% of the resting motor threshold (rMT) for the first dorsal interosseous of unaffected hemisphere.Two parts of Broca's area were sequentially stimulated: the anterior part (pars triangularis-PTr) and the posterior part (pars opercularis-POp). To target the regions of interest precisely, the coil was positioned on the scalp according to the coordinates used by Gough et al.The anterior stimulation site was 2.5 cm posterior to the canthus along the canthus-tragus line and 3 cm superior to this line; the posterior stimulation site was 4.5 cm posterior and 6 cm superior to the canthus-tragus line. The stimulation was applied in the same session with 1000 pulses over pars triangularis followed by 1000 pulses over pars opercularis in left hemisphere.All patients were evaluated before, after the end of last session of rTMS and after one month with ASRS and KAAT. The outcome measures were collected and statistically analyzed

ELIGIBILITY:
Inclusion Criteria:

* chronic post stroke nonfluent aphasia due to first-ever ischemic stroke in the distribution of middle cerebral artery diagnosed clinically and documented by computed tomography or magnetic resonance imaging on the brain
* Right handedness
* Both sexe groups
* Age ranged from 33 to 66 years old,
* Duration is at least 4 months from stroke onset,
* patients never received speech therapy before
* Educated for at least 10 years of education.

Exclusion Criteria:

* Aphasia due to head injury or neurological disease other than stroke,
* unstable cardiac dysrhythmia or cardiac pacemaker
* unstable or critically ill patients
* current or history of epilepsy, skull wounds and pregnant females.
* patients with severe grade of weakness which interfere with writing ability.

Ages: 33 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
evaluate the recovery of post stroke aphasia by non invasive procedure without language therapy | 1 month to assess the recovery
  rTMs is non invasive procedure may help improvement of speech performance

CONTACTS AND LOCATIONS:
Overall Officials: Haidy Elshebawy, lecturer, Principal Investigator — El kasr al ainy hospitals ,faculty of medicine ,cairo university
Locations (1):
- Haidy Elshebawy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fahmy EM, Elshebawy HM. Effect of High Frequency Transcranial Magnetic Stimulation on Recovery of Chronic Post-Stroke Aphasia. J Stroke Cerebrovasc Dis. 2021 Aug;30(8):105855. doi: 10.1016/j.jstrokecerebrovasdis.2021.105855. Epub 2021 May 25. PMID 34049013